CLINICAL TRIAL: NCT05584098
Title: Modified Early Warning Score (MEWS), Quick Sequential Organ Failure Assessment (qSOFA) and Physiological Parameters Combination to Predict the Occurrence of Sepsis in the Emergency Room
Brief Title: MEWS, qSOFA and Physiological Parameters Combination in the Emergency Room
Acronym: qSOFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Martin De Porress Hospital (Other)
Responsible Party: Principal Investigator, Chia-hsi Chen, attending physician,emergency medicine department, St. Martin De Porress Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21B-004
Record Dates: First submitted 2022-10-07; First posted 2022-10-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
Keywords: Sepsis; Modified Early Warning Score(MEWS); quick Sequential Organ Failure Assessment(qSOFA); emergency Medicine; physiological parameters combination
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: In a cross-sectional study, the investigator measures the outcome and the exposures in the study participants at the same time.
Masking Description: Mask all identified labels in all raw data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- qSOFA, MEWS and physiological parameters combination (Other): Modified Early Warning Score(MEWS), quick Sequential Organ Failure Assessment(qSOFA) and physiological parameters combination are used in prediction of occurrence of sepsis
  Interventions: Other: qSOFA, MEWS and physiological parameters combination

INTERVENTIONS:
Other: qSOFA, MEWS and physiological parameters combination — qSOFA ,MEWS and physiological parameters combination used in emergency medicine department could be helpful in the identification of the occurrence of sepsis

SUMMARY:
In the development of sepsis treatment of recent years, the demand for medical manpower has increased significantly when patients with sepsis appear because of the expansion of medical care demand and shortened response time related to sepsis Due to the shortage of manpower, a more simple and easy-to-operate inspection method is adopted and artificial intelligence technology is used to assist in the evaluation.

The applicability of physiological indicators MEWS, qSOFA and physiological parameters combination as sepsis screening tools in emergency department (ED) and predicting sepsis outcome in the emergency department. When patients with sepsis appear, artificial intelligence technology is used to remind the physicians to respond and administer drugs as soon as possible.

This is a single-center retrospective study of a group of patients admitted to the emergency department. The medical records were reviewed, mainly based on the hospital site records and the existing vital signs of the patients. Attended a hospital emergency room between January 2020 and December 2022. Physiological numerical indicators MEWS and qSOFA were all scored to understand the distribution of sepsis.

DETAILED DESCRIPTION:
1. A single-center retrospective study of a cohort of patients admitted to the emergency department
2. To see a doctor in the emergency department of the hospital between January 2020 and December 2022, review their medical records, and focus on the hospital's on-site records and the existing patient's vital signs.
3. The physiological indicators MEWS and qSOFA were scored to understand the distribution of sepsis.
4. Remind the doctor when a suspected sepsis patient appears under level 5 triage and use artificial intelligence technology to assist
5. This study will explore the specific improvement practices and effects of improving the response of patients with sepsis when they see a doctor
6. To analyze and evaluate the economics and benefits of this operation mode, improve the accuracy of emergency inspection of sepsis patients and improve the rationality of hospital manpower deployment
7. Scheduled progress of the plan: Patients who visited the emergency department of the hospital between January 2020 and December 2022 were included in this study under investigation. This is a retrospective study, and patients are required to undergo necessary examinations according to their own conditions, without any interference from the study

ELIGIBILITY:
Inclusion Criteria:

* This is a single-center retrospective study of a group of patients admitted to the emergency department.

Exclusion Criteria:

* Patients with incomplete treatment clinical data, lack of information in medical records, trauma patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
qSOFA used in emergency medicine department | From date of randomization until the date of first documented progression assessed up to 36 months
  The qSOFA score is a simple score consisting of three items: respiratory rate (RR) ≥ 22 breaths per minute, altered mentation (Glasgow Coma Scale [GCS] < 15), and systolic blood pressure (SBP) < 100 mmHg and lowest score is 1 and highest is 3. The more score will show more severe disease.
  MEWS score:Description Risk of death or ICU admission <3: patient in a stable condition, 3-4: Signs of respiratory failure. Consider higher level of care, ≥5: Patient in a critical condition. Higher level of care recommended
Modified Early Warning Score(MEWS) which quickly determine whether a particular patient needs increased medical attention | From date of randomization until the date of first documented progression assessed up to 36 months
  MEWS score = Systolic blood pressure + Heart rate + Urine output + Respiratory rate + Temperature + AVPU. The lowest score is 0 and highest score is 14. The more score will show more severe disease.
  MEWS score:Description Risk of death or ICU admission <3: patient in a stable condition, 3-4: Signs of respiratory failure. Consider higher level of care, ≥5: Patient in a critical condition. Higher level of care recommended
physiological parameters combination | From date of randomization until the date of first documented progression assessed up to 36 months
  Shock Index (SI) = Heart Rate / Systolic Blood Pressure Age-Adjusted Shock Index (Age SI) = Age x Shock Index Respiratory-Adjusted Shock Index (RASI) = HR/SBP × (RR/10)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsi Chen, MD, Principal Investigator — Emergency Medicine Department of St. Martin De Porres Hospital
Locations (1):
- St. Martin De Porres Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) is not available to other researchers